CLINICAL TRIAL: NCT04776551
Title: Percutaneous Trans-trapezial Fixation of Acute Scaphoid Fractures by Herbert Screw
Brief Title: Percutaneous Fixation of Acute Scaphoid Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Mohamed Mohamed Hamadouh, resident doctor, Sohag University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-21-2-09
Record Dates: First submitted 2021-02-14; First posted 2021-03-01 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Scaphoid Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group (1) (Other): group (1) who are complaining of acute scaphoid fractures,we will do percutaneous trans trapezial fixation of scaphoid by Herbert screw.Short arm circular cast including the thumb will be applied. After 3 weeks, cast will be removed and exercises will start.
  Interventions: Procedure: Percutaneous fixation of acute Scaphoid fractures

INTERVENTIONS:
Procedure: Percutaneous fixation of acute Scaphoid fractures — Percutaneous Trans-trapezial fixation of acute Scaphoid fractures by Herbert screw

SUMMARY:
Percutaneous Trans-trapezial fixation of acute Scaphoid fractures by Herbert screw

DETAILED DESCRIPTION:
Aim of the work:

To assessment outcomes of percutaneous Trans-trapezial fixation of acute scaphoid fracture.

Operative Technique:

Anesthesia: carried out under general anesthesia or brachial plexus block and under tourniquet control.

Position: supine. Approach: Percutaneous Trans-trapezial fixation of acute Scaphoid fracture. Recording any intraoperative complication that may affect the result.

Postoperative Follow Up:

Short arm circular cast including the thumb will be applied. After 3 weeks, cast will be removed and exercises will start.

ELIGIBILITY:
Inclusion Criteria:

* - Acute stable non displaced waist fracture (A2).
* Acute unstable oblique distal third (B1).
* Acute unstable displaced waist (B2).
* Acute un stable fracture dislocation (B4).
* Acute un stable comminuted fracture (B5).

Exclusion Criteria:

* - Acute stable fracture tubercle (A1).
* Acute unstable fracture proximal pole (B3).
* Delayed union fracture (C).
* Established non-union fracture includes fibrous (D1) and sclerotic (D2).
* Bilateral fractures because of possible interference with postoperative grip strength measurement.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change of wrist power | Up to 18 months
  Modified Mayo wrist score

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospital, Sohag, Egypt